CLINICAL TRIAL: NCT03772977
Title: The Brain Health Champion Study: Promoting Non-pharmacological Interventions in Cognitive Disorders and Those at Risk
Brief Title: The Brain Health Champion Study
Acronym: BHC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Seth Gale, Associate Neurologist, Assistant Professor of Neurology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000384
Record Dates: First submitted 2018-11-25; First posted 2018-12-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment; Dementia, Mild; Subjective Cognitive Decline; At Risk for Cognitive Decline
Keywords: mild cognitive impairment; dementia risk reduction; brain health
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Health Champion (BHC) (Experimental): A "health coach" intervention with weekly phone calls
  Interventions: Behavioral: Brain Health Champion
- Standard of Care (SOC) (No Intervention): The current physician/provider counseling on brain health to reduce cognitive decline or incidence of cognitive impairment that occurs, per providers' own practice

INTERVENTIONS:
Behavioral: Brain Health Champion — A health coach embedded within an existing clinical care team
  Arms: Brain Health Champion (BHC)

SUMMARY:
6-month, randomized, controlled investigation measuring the effect of increased clinical contact and personalization compared to standard physician counseling on adherence to consensus-based, brain health recommendations for patients with subjective cognitive decline, mild cognitive impairment, and early dementia or patients who are at risk for developing these conditions.

DETAILED DESCRIPTION:
This is a 6-month, randomized, controlled investigation measuring the effect of increased clinical contact and personalized recommendations from a health coach, compared to standard physician counseling on adherence to consensus-based, brain health recommendations, including 80 patients with either subjective cognitive decline, MCI, or early dementia enrolled from a hospital-based memory disorders clinic, or, with risk factors for dementia enrolled from a hospital-based primary care clinic. Participants and caregivers in the health coach arm work with a health coach within their respective practice, called the a "brain health champion" (BHC), through weekly motivational phone calls every 6 weeks. In the encounters and visits, BHCs and patients/caregivers work together to establish, update, and achieve personalized, attainable lifestyle goals. Participants in the control arm receive standard counseling and education from providers during routine clinic visits. Changes in physical activity, dietary pattern, and social and cognitive activities are measured using questionnaires validated in cognitively impaired and normal populations. Other outcomes include measures of quality of life (QOL), cognitive function, neuropsychiatric status, sleep quality, and behavior. Follow-up assessments are also completed at 6 months post-intervention, with some patients receiving "booster" encounters to assess the maintenance of behaviors.

ELIGIBILITY:
Inclusion criteria:

* Be age 60 to 79
* Existing patient at Brigham Health system with at least one prior visit with providers and plans to establish/continue longitudinal care
* Be sufficiently fluent in the English language to understand instructions and perform the cognitive and functional tests
* For neurology participants only: Have a diagnosis of Subjective Cognitive Disorder (SCD) (MMSE guideline 27-30), Mild Cognitive Impairment (MCI) due to Alzheimer disease (AD), cerebrovascular disease (CVD), or mixed-type AD/CVD (MMSE guideline 24-30), or mild dementia due to AD, CVD, or mixed-AD/CVD (MMSE guideline 20-30). In some cases, based on the clinical judgment of the treating neurologist, we may enroll a patient who falls outside of these guidelines or whose diagnosis and overall level of functioning does not perfectly correlate to their MMSE score.
* For primary care participants only: Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) dementia risk score of ≥ 6, or score of 5 plus one of the following: a history of ADRD in a first-degree relative, or type II diabetes or "pre-diabetes" spectrum (A1C level ≥ 5.7)

Exclusion criteria:

* Be enrolled in another health behavior or non-pharmacologic intervention for a neurocognitive disorder
* Be unable to or unwilling to carry out regular physical exercise, multiple times weekly.
* Be not recommended to participate by their Internist/Primary Care Provider due to health-related concerns.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-report adherence to Mediterranean diet | 6 months
  Goulet Mediterranean Diet Score (questionnaire).
  Measured adherence to the Mediterranean Diet. Likert Scale 0-44, with higher values indicating stronger adherence to the dietary pattern.
Self-report participation in cognitive and socially stimulating activities | 6 months
  Florida Cognitive Activities Scale (questionnaire).
  Measures participation in socially and cognitively stimulating activities. Likert Scale 0-180, with higher values indicating greater participation.
Self-report exercise and physical activity | 6 months
  Physical Activity Scale for the Elderly (questionnaire).
  Measures walking, moderate, and vigorous activity. Zero lower limit, no upper limit. Higher values indicate more physical activity.

SECONDARY OUTCOMES:
Quality of Life Self-Report | 6 months
  Flanagan Quality of Life Scale (questionnaire).
  Measures quality of life. Likert scale 0-112, higher values indicate higher quality of life.
Neuropsychiatric status | 6 months
  Neuropsychiatric Inventory Questionnaire.
  Measures caregiver report of 12 neuropsychiatric symptoms, severity (1-3) and distress (0-5) with higher values indicating more neuropsychiatric symptoms.
Cognitive function | 6 months
  Mini Mental Status Examination: Multidomain cognitive test, scored 0-30.
  PACC-BHC: Neurosychological test battery including: 1) Free and Cued Selective Reminding Test (FCSRT); 2) Logical Memory, immediate and delayed Story Recall; 3) Visual Paired Associates; 4) Digit-Symbol Substitution Test; 5) Trail Making Test, Part A; 6) Trail Making, Part B; 7) Number Span, 8) Category Fluency (animals, fruits, vegetables); and 9) Phonemic Fluency.
Sleep | 6 months
  Medical Outcomes Study Sleep Scale
  Likert scale measuring sleep quality and sleep problems index. 0-60 with greater values representing higher sleep quality and lower sleep problems.

CONTACTS AND LOCATIONS:
Overall Officials: Seth A Gale, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Department of Neurology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz HEM, Bay CP, McFeeley BM, Krivanek TJ, Daffner KR, Gale SA. The Brain Health Champion study: Health coaching changes behaviors in patients with cognitive impairment. Alzheimers Dement (N Y). 2019 Nov 12;5:771-779. doi: 10.1016/j.trci.2019.09.008. eCollection 2019. PMID 31763431
- See also: Related Info — https://brainhealth.bwh.harvard.edu/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT03772977/Prot_SAP_001.pdf